CLINICAL TRIAL: NCT02737371
Title: F901318 - A Phase I, Double-Blind, Placebo Controlled, Multiple Ascending Oral Dose Safety, Tolerability and Pharmacokinetic Study in Healthy Male and Female Subjects
Brief Title: Multiple Ascending Oral Dose Study of F901318 in Healthy Subjects
Acronym: ORALMAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: F2G Biotech GmbH (Industry)
Collaborators: SimbecRresearch Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F901318-01-06-16
Record Dates: First submitted 2016-03-23; First posted 2016-04-13 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Invasive Aspergillosis
MeSH Terms: interventions — Antifungal Agents

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- F901318 Dose level A oral (Experimental): F901318 adverse events days 1-10
  Interventions: Drug: F901318 Dose level A oral
- Placebo Dose level A oral (Placebo Comparator): Placebo adverse events days 1-10
  Interventions: Drug: Placebo dose level A oral
- F901318 Dose level B oral (Experimental): F901318 adverse events days 1-10
  Interventions: Drug: F901318 Dose level B oral
- Placebo Dose level B oral (Placebo Comparator): Placebo adverse events days 1-10
  Interventions: Drug: Placebo dose level B oral
- F901318 Dose level C oral (Experimental): F901318 adverse events days 1-10
  Interventions: Drug: F901318 Dose level C oral
- Placebo Dose level C oral (Placebo Comparator): Placebo adverse events days 1-10
  Interventions: Drug: Placebo Dose level C oral

INTERVENTIONS:
Drug: F901318 Dose level A oral — Adverse events days 1-10
  Other Names: antifungal agent
  Arms: F901318 Dose level A oral
Drug: Placebo dose level A oral — Placebo adverse events days 1-10
  Arms: Placebo Dose level A oral
Drug: F901318 Dose level B oral — F901318 adverse events days 1-10
  Other Names: antifungal agent
  Arms: F901318 Dose level B oral
Drug: Placebo dose level B oral — Placebo adverse events days 1-10
  Arms: Placebo Dose level B oral
Drug: F901318 Dose level C oral — F901318 adverse events days 1-10
  Other Names: antifungal agent
  Arms: F901318 Dose level C oral
Drug: Placebo Dose level C oral — Placebo adverse events days 1-10
  Arms: Placebo Dose level C oral

SUMMARY:
Double blind, placebo controlled, ascending multiple (10) oral dose, sequential group study. Twenty-four subjects will complete the study in 3 cohorts (Groups A to C), each group consisting of 8 subjects. Each cohort will consist of 4 male and 4 female subjects. Each subject will be dosed for 10 days and will be on study for approximately 7 weeks. Each subject will participate in one treatment cohort only, residing at the Clinical Research Unit (CRU) from Day -1 (the day before dosing) to Day 15 (120 hours post the last dose). The dose will range between 2 and 10 mg/kg daily, given as either a single daily dose or as two doses divided over the 24-hour dosing period.

All subjects will return for a post-study visit 8 to 10 days after the last dose of study medication.

Cohorts will be dosed at least at 3 weekly intervals. There will be a review of the safety and pharmacokinetic data of each cohort prior to each dose escalation.

DETAILED DESCRIPTION:
Male and female healthy subjects conforming to the selection criteria will be invited to take part in the study.

Screening visit (Visit 1) After giving fully informed, written consent, subjects will attend the clinic.

Subjects will undergo screening within 28 days prior to the first dose administration. Prior to the screening visit, subjects will:

* Refrain from vigorous exercise for 7 days
* Abstain from alcohol for 48 hours
* Subjects will sign the consent form in the presence of a CRU physician prior to any screening procedures being performed. The information recorded for all subjects, regardless of their suitability for the study, will be retained and archived.

The following information and procedures will be recorded and performed as part of the screening assessments:

* Medical history
* Ethnic origin, sex, age, height, weight, and BMI
* Vital signs: supine blood pressure, supine pulse rate, and oral body temperature
* Resting 12 lead ECG
* Physical examination
* Urine drugs of abuse screen, cotinine and alcohol breath test
* Pregnancy test, which must be negative
* Fasting clinical laboratory and serology investigations
* All females will be asked to give the approximate date of the last menstrual period.
* Ophthalmological assessments (Performed at a second screening visit in subjects who have been shown at the first screening visit to meet eligibility criteria for the study)

Up to 28 days after screening, subjects will attend the clinic. Subjects will be admitted to the research unit at approximately 09:00 hours in the morning the day before dosing (Day -1). Urine will be subjected to a screen for drugs of abuse and detection of any of these substances which will disqualify the subject from the study. A physical examination, check of inclusion/exclusion criteria, clinical laboratory evaluations, pregnancy test where relevant and which must be negative, oral temperature and body weight will be performed. Subjects will be asked whether they have experienced any adverse events or taken any concomitant medication since their previous visit. Supper will be served starting at approximately 19.30 hours and a snack at approximately 21.00 hours after which they will fast overnight and until 4 hours post dose. Water will be allowed ad libitum throughout.

On Day 1, the total first urine void of the morning for each subject will be collected into a polyethylene container and, from this, a sample will be taken for urinalysis and pre-dose / baseline F901318 concentration. Within one hour before dosing commences ( 1 hour), blood will be drawn for laboratory safety assessments (haematology and clinical chemistry), and pre-dose baseline F901318 and metabolites concentration. Supine and standing blood pressure and pulse rate in duplicate, body temperature and a 12-lead ECG will be recorded. The subjects will also be connected to continuous ECG recording from -1 hour) until at least 12 hours after the start of dosing.

Subjects will be asked whether they have experienced any adverse events overnight. Any concomitant medications will be recorded.

Subjects will then be dosed. This will be an oral suspension washed down with 250 mL of phosphate buffer. Subjects will be dosed with regular intervals between each subject.

After dosing, the following measurements and observations will be obtained:

* Blood samples for analysis of F901318 plasma concentration will be drawn at 15min, 30 min, 45min, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12 and 16 hours after dosing on Day 1.
* On Days 2 to 9, pharmacokinetic blood samples will be drawn within 15 minutes prior to dosing and 2 and 4 hours later.
* On Day 10, blood samples for pharmacokinetic analysis will be drawn within 15 minutes of the commencement of dosing and 15min, 30 min, 45min,1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96 and 120 hours following dosing.
* Pharmacokinetic blood samples will be analysed and reviewed before each dose escalation. After the first dose level administration, the dose level and the timing of each blood sample may be adjusted for the subsequent dose escalation. The basis for this decision will depend upon the pharmacokinetic profiles obtained from the preceding group of subjects. All changes will be documented in a file note. The number of samples or volume of blood drawn must not be increased without prior approval of the relevant ethics committee.
* If it appears that Cmax may exceed the stopping criteria, the daily dose for that cohort will be divided into to two halves given 6-12 hours apart with the exception of Day 10 on which a single morning half dose will be given. The changes will be made on the basis of pharmacokinetic predictions using data obtained from previous cohorts. In that case, blood and urine sampling times will be adjusted accordingly and documented in a note to file. The number of blood samples drawn for pharmacokinetics will not exceed 68 without approval of the relevant ethics committee.
* Blood samples will be drawn for metabolite measurements 4 and 8 hours after the morning dose on Day 1 and within 15 minutes prior to and 4 and 8 hours after the dose on Day 10.
* Blood will be collected for safety measurements (haematology and clinical chemistry) and a urine sample will be obtained for urinalysis on Days 2, 3, 4, 5, 6, 7, 8 and 9 in the 15 minutes prior to the morning dose and 24, 48 and 72 hours after the dose on Day 10.
* Complete urine collections for analysis of F901318 urine concentration will be made for the following intervals in relation to dosing: 0-4, 4-8, 8-12, 12-24 hours on Day 1 and 0-4, 4-8, 8-12, 12-16, 16-24, 24-48, 48-72, 72-96 and 96-120 hours after the dose on Day 10.
* Supine and standing pulse rate and blood pressure and body temperature (vital signs) will be recorded 30, 60 and 120 minutes, 4, 8 and 12 hours after dosing on Day 1, prior to (within 30 minutes) dosing on Days 2 - 10 and 4 hours after dosing on Days 2 - 10.
* Twelve-lead ECGs will be obtained 1, 4, 8, and 12 hours after dosing on Day 1 and within 30 minutes before and 4 hours after dosing on Days 3, 6 and 10.
* The continuous ECG recording will cease 12 hours after dosing on Day 1. It may be extended to 24 hours at the discretion of the PI. A further continuous recording will be obtained from one hour prior to and for 12 hours after the dose on Day 10. It also may be extended to 24 hours at the discretion of the PI.
* Spontaneously reported adverse events and concomitant medications will be noted throughout.
* Lunch will be served approximately 4 hours after each morning dose but after all the 4 hour observations and blood sampling have been completed and a main meal will be served approximately 8 hours and a snack approximately 11.5 hours after each morning dose.
* Ophthalmological evaluation will be conducted 24 hours post Day 10 dosing (+/- 4 hours)
* A pregnancy test will be performed on Day 15 in females of child bearing potential.

Subjects may leave the Research Unit on Day 15, unless they have experienced adverse events that, in the opinion of the Investigator, warrant further observation and/or treatment.

All subjects will be followed up 8-10 days after the last dose of study drug with a post-study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be males or females of any ethnic origin between 18 and 45 years of age and with a body weight of 50-100 kg inclusive. Females of child bearing potential must be established on a reliable form of contraception and have a negative pregnancy test at screening.
2. Subjects must be in good health, as determined by a medical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations (congenital non haemolytic hyperbilirubinaemia is acceptable).
3. Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions.
4. Subjects must have ophthalmology assessments within the normal limits at screening. This includes normal Meibomian gland function.

Exclusion Criteria:

1. Male or female subjects who are not willing to use appropriate contraception during the study and until 3 months after the last dose.
2. Subjects who have received any prescribed systemic or topical medication within 14 days of the dose administration unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety.
3. Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days of the dose administration (with the exception of vitamin/mineral supplements and paracetamol) unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety.
4. Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of the dose administration unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety.
5. Subjects who are still participating in a clinical study (e.g. attending follow-up visits) or who have participated in a clinical study involving administration of an investigational drug (new chemical or biological entity) in the past 3 months since the last dose.
6. Subjects who have donated any blood, plasma or platelets in the 3 months prior to screening or who have made donations on more than two occasions within the 12 months preceding the dose administration.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-05-22 (Actual); Study Completion 2017-05-22 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability | 10 days
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability

SECONDARY OUTCOMES:
Pharmacokinetics Area under concentration/time curve | 15 days
  Area under concentration/time curve

CONTACTS AND LOCATIONS:
Overall Officials: Girish Sharma, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research Ltd, Merthyr Tydfil, Glamorgan, United Kingdom

IPD SHARING:
Plan to Share IPD: No